CLINICAL TRIAL: NCT01548495
Title: Investigating Recombinant Human Erythropoietin (rHuEPO) Treatment Efficacy Depending on the Presence of Erythropoietin Autoantibodies in Myelodysplatic Syndrome (MDS) Patients
Brief Title: Autoantibodies Against Human Recombinant Erythropoietin in Myelodysplatic Syndrome Patients
Acronym: MDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: yair levy (Other)
Responsible Party: Sponsor-Investigator, yair levy, director of internal medicin E department, Meir Medical Center
Organization: Meir Medical Center (Other)
Other Study IDs: MDS-2011
Record Dates: First submitted 2012-02-28; First posted 2012-03-08 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Myelodysplatic Syndrome
Keywords: MDS; Autoantibodies; Erythropoietin; Autoantibodies in MDS patients treated with EPO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Responded to rHuEPO treatment: response to EPO was defined as a rise in untransfused hemoglobin concentration of at least 2 g/dl or a 50% decrease in transfusion requirements over the treatment period
- IR to rHuEPO treatment: No rise in hemoglobine consentration at normal and high dose rHuEPO treatment
- Responded to high level rHuEPO: Responded to more than 80,000UI of rHuEPO treatment
- No rHuEPO treatment

SUMMARY:
The purpose of this study is to verify the presents of autoantibodies in serums of MDS serum patients who had an inadequate response or did not respond to Recombinant human erythropoietin (rHuEPO) treatment.

DETAILED DESCRIPTION:
MDS are a heterogeneous group of hematologic disorders broadly characterized by cytopenias associated with a dimorphic and usually cellular bone marrow, and by consequent ineffective blood cell production. 85% of patients have a severe anemia which is Associated with lowering quality of life and Often requires blood transfusions. Historically, only stem cell transplantation offers cure. however, multiple new drugs have been approved for treatment, such as to Recombinant human erythropoietin (rHuEPO) treatment for dealing with the anemia. rHuEPO treatment can improve hematocrit level in 25% of patient which leaves the rest with the need of other treatment solution. Studies have shown presents of anti- rHuEPO in blood serums which followed Treatment of other diseases. These findings can indicate the possibility of the presence of antibodies in MDS patients as well.

ELIGIBILITY:
Inclusion Criteria:

* Followed up hematological patients
* Pateint recieving rHuEPO treatment (except control group)
* Pateint signed informed consent

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDS patient from meir health care center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Correlate the Presence of Erythropoietin autoantibodies titer in MDS patients with an inadequate response (IR) to Human Recombinant Erythropoietin treatment | 1 year
  Response to Erythropoietine (EPO) was defined as a rise in untransfused hemoglobin concentration of at least 2 g/dl or a 50% decrease in transfusion requirements over the treatment period.
  Detection of Erythropoietin autoantibodies was performed by "Home-made ELISA" test.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical center, Kfar Saba, Israel, Israel